CLINICAL TRIAL: NCT02844660
Title: A Multicenter, Prospective, Randomized, Controlled, Comparative Parallel Study of Dehydrated Human Umbilical Cord Allograft in the Management of Diabetic Foot Ulcers
Brief Title: Dehydrated Human Umbilical Cord Allograft in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECDFU001
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes Mellitus; Foot Diseases; Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Diseases; Foot Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EpiCord (Experimental): Weekly application of EpiCord and standard of care (moist wound therapy and offloading)
  Interventions: Biological: EpiCord
- Standard of Care (Active Comparator): Weekly application of moist wound therapy and offloading
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: EpiCord — Weekly application of EpiCord and standard of care (moist wound therapy and offloading)
  Arms: EpiCord
Other: Standard of Care — moist wound therapy and offloading
  Arms: Standard of Care

SUMMARY:
A Multicenter, Prospective, Randomized Controlled Comparative Parallel Study To determine the safety and effectiveness of EpiCord as compared to standard of care (SOC) therapy for the treatment of chronic, non-healing diabetic foot ulcers (DFUs)

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial. The trial will include approximately 66 subjects in up to 10 experienced clinical centers in the United States. The estimated enrollment period is 18 weeks (this includes the 2-week run-in period). After completing a 2-week screening period, the subjects will be followed for at least 16 weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a known history of Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).

2. Index ulcer characteristics:

a. Ulcer present for ≥ 30 days prior to randomization (Day 0) b. Index ulcer is located below the ankle c. Index ulcer area after debridement is ≥ 1 cm² and ≤ 15 cm² at the randomization visit 3. Subject has completed 14-day run-in period with ≤ 30% wound area reduction post-debridement.

4. Subject has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

* Dorsum transcutaneous oxygen test (TcPO2) with results ≥ 30 mmHg, OR
* ABIs with results of ≥ 0.7 and ≤ 1.2, OR
* Doppler arterial waveforms, which are triphasic or biphasic at the ankle of the affected foot 5. Age ≥ 18 6. The subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study

  1. Index Ulcer Assessment:

     1. Penetrates down totendon, or bone
     2. Presence of another diabetic foot ulcer within 3 cm of the index ulcer
     3. Index ulcer determined to be due to active Charcot deformity or major structural abnormalities of the foot
     4. Exhibits clinical signs and symptoms of infection
     5. Known or suspected local skin malignancy to the index diabetic ulcer
     6. Wound duration > one year without intermittent closure
  2. Prior therapies - Subjects receiving treatment with any of the following will not be eligible for enrollment:

     1. In the last 7 days - Negative pressure wound therapy (wound vac or SNaP®) of the index ulcer
     2. In the last 7 days - Hyperbaric oxygen (HBO) therapy
     3. In the last 10 days - Chemical debridement, Dakin's solution, medical honey therapy
     4. In the last 30 days - Treatment with cytotoxic chemotherapy, application of topical steroids to the ulcer surface, or use of ≥ 14 days of immune-suppressants (including systemic corticosteroids); or, subject is anticipated to require such medications during the course of the study
     5. In the last 30 days - study ulcer treatment with any biological skin substitutes, including EpiCord, biomedical or topical growth factors, tissue engineered materials (e.g. Apligraf® or Dermagraft®), or other scaffold materials (e.g. OASIS® Wound Matrix, MatriStem® Wound Matrix, Grafix, etc.)
     6. In the last 30 days - Subject has been on any investigational drug(s) or therapeutic device(s)
     7. In the last 6 months - Amputation or revascularization (surgical or stenting) to the affected leg or foot
  3. Subject criteria that will make subject ineligible for enrollment:

     1. Known osteomyelitis or active cellulitis at wound site
     2. Hemoglobin A1C >12 in the last 60 days prior to randomization
     3. History of Immune system disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or HIV
     4. Allergy or known sensitivity to Aminoglycosides such as gentamicin sulfate and/or streptomycin sulfate
     5. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator
     6. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
     7. Known history of poor compliance with medical treatments
     8. Subjects currently enrolled in this study. Concurrent enrollment in the study is prohibited
     9. Subjects currently receiving radiation therapy or chemotherapy
     10. Patients currently on dialysis or planning to start dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Complete Ulcer Closure | 12 weeks
  The percentage of subjects with complete closure of the study ulcer as assessed by photographic evaluation
Study Safety Measurement | 12 weeks
  The proportion of product related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events at 12 weeks.

SECONDARY OUTCOMES:
Time to complete closure | up to 12 weeks
  As assessed by photographic evaluation and the Investigator
Rate of wound closure | up to 12 weeks
  As assessed by photographic evaluation and the Investigator
Incidence of ulcer recurrence | up to 12 weeks
  Incidence of ulcer recurrence at the site of the study ulcer
Quality of Life Health Survey | up to 12 weeks
  Change in quality of life metrics as measured by SF-36 Health Survey
Quality of Life-Pain | up to 12 weeks
  Change in quality of life metrics as measured by changes in the patients reported pain scores as measure by the Visual Analog Scale
Cost effectiveness of treatment | up to 12 weeks
  Cost effectiveness of treatment regime. looking at the number of grafts used on each study subject throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: William Tettelbach, MD, Principal Investigator — Intermountain Medical Center
Locations (13):
- United States (13):
  - Central Research Associates, Birmingham, Alabama
  - Arizona Regional Medical Research (ARMR), Tucson, Arizona
  - ILD Research, Carlsbad, California
  - Limb Preservation Platform, Inc, Fresno, California
  - Foot and ankle clinic, Los Angeles, California
  - Doctors Research Network, Miami, Florida
  - Joseph M. Still Burn Center at Doctors Hospital, Augusta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Foot and Ankle Center, Haverford, Pennsylvania
  - Futuro Clinical Trials, McAllen, Texas
  - Ambulatory Foot & Ankle Center, PC, Hampton, Virginia
  - Costal Podiatry, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No